CLINICAL TRIAL: NCT04829747
Title: A Phase 3, Multicenter, Open-Label, 12-Week Study to Evaluate the Safety and Tolerability of Oral Atogepant for the Prevention of Migraine in Chinese Participants With Chronic Migraine
Brief Title: Study to Assess Adverse Events (AEs) When Oral Atogepant Tablet is Given to Adult Chinese Participants Who Completed Study 3101-303-002 to Prevent Chronic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3101-311-002
Record Dates: First submitted 2021-04-01; First posted 2021-04-02 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Chronic Migraine
Keywords: Chronic Migraine; Migraine; Atogepant; AGN-241689
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atogepant (Experimental): Participants will receive fixed dose of Atogepant once daily for 12 weeks.
  Interventions: Drug: Atogepant

INTERVENTIONS:
Drug: Atogepant — Oral Tablet

SUMMARY:
Migraine is characterized by attacks of throbbing, moderate or severe headache, associated with nausea, vomiting, and/or sensitivity to light and sound. The main objective of the study is to evaluate how safe and effective the atogepant is in preventing chronic migraine in adult Chinese participants who completed study 3101-303-002. Adverse events will be monitored.

Atogepant is an investigational drug being developed to prevent chronic migraine. All participants will receive the same treatment. Approximately 120 adult participants who completed study 3101-303-002 will be enrolled at approximately 25 centers in China.

All participants will receive atogepant oral tablet once daily for 12 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants completed the double-blind treatment period, and the safety follow-up period, if applicable, depending on the timing of study initiation, of Study 3101-303-002 without significant protocol deviations and who did not experience an adverse event (AE) that, in the investigator's opinion, may indicate an unacceptable safety risk.

Exclusion Criteria:

* Participants requiring any medication, diet, or nonpharmacological treatment on the list of prohibited concomitant medications or treatments, that cannot be discontinued or switched to an allowable alternative. Concomitant medications with demonstrated efficacy for the prevention of migraine is exclusionary, except that participants from lead-in study 3101-303-002 taking 1 medication with demonstrated efficacy for the prevention of migraine may participate in the current study provided that the dose was stable prior to the lead-in study and the participant is willing to continue taking that medication.
* Participants with an electrocardiogram (ECG) indicating clinically significant abnormalities at Visit 1.
* Participants with hypertension (sitting systolic blood pressure (BP) > 160 mm Hg or sitting diastolic BP > 100 mm Hg) at Visit 1.
* Participants with a significant risk of self-harm Columbia-Suicide Severity Rating Scale (C-SSRS), or of harm to others (investigator opinion); participants who report suicidal ideation with intent, with or without a plan, since the last visit, must be excluded.
* Participants with clinically significant hematologic, endocrine, cardiovascular, pulmonary, renal, hepatic, gastrointestinal, or neurologic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (3):
- China (3):
  - Chinese PLA General Hospital /ID# 227546, Beijing, Beijing Municipality
  - The Second Hospital of Shanxi Medical University /ID# 227567, Taiyuan, Shanxi
  - The second Affiliated hospital of Zhejiang University school of Medicine /ID# 227558, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2 subjects were included in the modified intent-to-treat (mITT) population, defined as all subjects who received ≥1 dose of study treatment (atogepant) in this extension study and had ≥1 evaluable postbaseline 4-week period of electronic diary (eDiary) data in this extension study. A total of 3 subjects were included in the safety population, defined as all subjects who received ≥1 dose of the study treatment (atogepant) in this extension study.
Period: Overall Study
Arm/Group | Atogepant
Started | 3
Completed | 2
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: The safety population, consisting of all participants who received at least 1 dose of study intervention (atogepant) in this extension study.
Arm/Group | Atogepant
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  Years of Age: 33 Years Old | 1
  Years of Age: 41 Years Old | 1
  Years of Age: 51 Years Old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity.
Time Frame: Baseline of the study 3101-303-002 to 16 weeks
Population: Safety population: all subjects who received ≥1 dose of the study treatment (atogepant) in this extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Atogepant
Number analyzed (Participants) | 3
Participants | 1

2. Primary Outcome: Number of Participants With Significant Change in Clinical Laboratory Determinations
Description: Number of participants with clinically significant change from baseline for any detectable clinical laboratory tests like hematology will be reported.
Time Frame: Baseline of the study 3101-303-002 to 16 weeks
Population: Safety population: all subjects who received ≥1 dose of the study treatment (atogepant) in this extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Atogepant
Number analyzed (Participants) | 3
Participants | 0

3. Primary Outcome: Number of Participants With Significant Change in Vital Sign Measurements
Description: Number of participants with clinically significant change from baseline for any vital signs like standing BP, sitting and standing pulse rate will be reported.
Time Frame: Baseline of the study 3101-303-002 to 16 weeks
Population: Safety population: all subjects who received ≥1 dose of the study treatment (atogepant) in this extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Atogepant
Number analyzed (Participants) | 3
Participants | 0

4. Primary Outcome: Number of Participants With Significant Change in Electrocardiogram (ECG) Parameters
Description: 12-lead ECG will be performed.
Time Frame: Baseline of the study 3101-303-002 to 12 weeks
Population: Safety population: all subjects who received ≥1 dose of the study treatment (atogepant) in this extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Atogepant
Number analyzed (Participants) | 3
Participants | 0

5. Primary Outcome: Number of Participants With a Change in Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior. Suicidal ideation is classified on a 5-item scale: 1 being wish to be dead and 5 being active suicidal ideation with specific plan and intent. Suicidal behavior is classified on a 5-item scale: 0 being no suicidal behavior and 4 being actual attempt.
Time Frame: Baseline of the study 3101-303-002 to 16 weeks
Population: Safety population: all subjects who received ≥1 dose of the study treatment (atogepant) in this extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Atogepant
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 16 Weeks
Description: An AE was considered a treatment-emergent adverse event (TEAE) if it began or worsened (increased in severity or became serious) on or after the date of the first dose of double-blind study treatment in the lead-in study. TEAEs could have been identified as those AEs captured in this study with recorded onset date on or after the date of the first dose of lead-in double-blind study treatment and within 30 days after the last dose of open-label study treatment or Visit 5, whichever came later.
Arm/Group | Atogepant
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atogepant (N=3)
DYSMENORRHEA (Reproductive system and breast disorders) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT04829747/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT04829747/SAP_001.pdf